CLINICAL TRIAL: NCT04229550
Title: Metabolic Effects of One-Week Heavy Drinking and Fast Food Intake During Roskilde Festival in Young Healthy Male Adults
Brief Title: Metabolic Effects of One-weak Heavy Drinking
Acronym: ROSMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-15019685
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Metabolic Disturbance; Alcohol; Harmful Use; Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control subjects (No Intervention): 1 week of normal daily life and only by the National Health Board recommendated alcohol consumption.
- Festival subjects (Experimental): 1 week's participation in Roskilde Festival 2016
  Interventions: Behavioral: Festival participation

INTERVENTIONS:
Behavioral: Festival participation — One week's participation in Roskilde Festival 2016 or living a normal daily life.
  Arms: Festival subjects

SUMMARY:
Examination of the effect of one week's unhealthy lifestyle on glucose metabolism and liver parameters in a group of young, healthy males participating in Roskilde Festival 2016.

DETAILED DESCRIPTION:
Metabolic effects of intermittent unhealthy lifestyle in otherwise young healthy adults are poorly studied. The investigators evaluated the effect of one week's unhealthy lifestyle on glucose metabolism and liver parameters in a group of young, healthy males participating in Roskilde Festival 2016.

Festival participants were studied before and after participation (one week) in Roskilde Festival 2016 and matched with controls who lead a normal life for an equivalent period of time. An oral glucose tolerance test (OGTT), abdominal ultrasound and strain elastography for liver stiffness were performed together with a bioimpedance scan and cognitive tests.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18,5-25 kg/m2
* Normal liver function (assessed by ASAT, ALAT, GGT, alkaline phosphatase, albumin and bilirubin, coagulation factors II, VII and X, INR and platelets)

Exclusion Criteria:

* Planning alcohol withdrawal or dieting/a special low-fat diet during Roskilde Festival
* Diabetes or pre-diabetes
* First degree relatives with diabetes
* Kidney disease (eGFT<60 ml/min and/or albuminuria)
* Chronic diseases (in addition to those already mentioned) that could affect participation in festival activities (concerts and parties)
* Any condition in which the investigator believed would make it impossible to participate

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-07-04 (Actual); Study Completion 2016-07-04 (Actual)

PRIMARY OUTCOMES:
Impairment of glucose tolerance | First day after intervention week
  Evaluated by OGTT

SECONDARY OUTCOMES:
Hepatic steatosis | First day after intervention week
  Evaluated by abdominal ultrasound scan

OTHER OUTCOMES:
Altered cognitive function | First day after intervention week
  Evaluated by validated cognitive test ("SCIP")

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, Prof,MD,PhD, Principal Investigator — University of Copenhagen

IPD SHARING:
Plan to Share IPD: No